CLINICAL TRIAL: NCT05570474
Title: Effect of Protein Supplementation on Fat Free Mass Preservation After Bariatric Surgery, a Randomized Double-blind Placebo-controlled Trial.
Brief Title: Effect of Protein Supplementation on Fat Free Mass Preservation After Bariatric Surgery
Acronym: PROMISE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maasstad Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: L2022059
Record Dates: First submitted 2022-09-26; First posted 2022-10-06 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Bariatric Surgery Candidate; Protein Deficiency; Muscle Loss
Keywords: bariatric surgery; RYGB; Roux-en-Y gastric bypass; protein supplementation; fat free mass; muscle mass
MeSH Terms: conditions — Protein Deficiency; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated to either protein group or placebo group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study products (protein or placebo drinks) are provided to study participants. Study product is marked by a unique batch number, corresponding to protein or placebo in the ingredients list.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protein (Experimental): Daily protein shake during 6 months after surgery
  Interventions: Dietary Supplement: Protein drink supplementation
- Control (Placebo Comparator): Daily placebo shake during 6 months after surgery
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Protein drink supplementation — Daily drink containing 20 grams of whey protein, dissolved in 200mL water.
  Arms: Protein
Dietary Supplement: Placebo — Daily placebo drink
  Arms: Control

SUMMARY:
This double blind randomized placebo controlled trial investigates the effect of protein supplementation on fat free mass loss in patients who underwent a Roux-en-Y gastric bypass.

DETAILED DESCRIPTION:
Rationale: Protein malnutrition is a severe complication of bariatric surgery and leads to increased morbidity. Previous studies have shown that protein intake and physical activity are the most important factors in the preservation of fat free mass during weight loss. Low protein intake is very common in patients undergoing bariatric surgery despite dietary counselling. Protein powder supplements might help patients to achieve the protein intake recommendations after bariatric surgery and could therefore contribute to preserve fat free mass.

Objective: The main aim of this study is to assess the effect of a daily consumed clear protein powder shake during the first six months after bariatric surgery on fat free mass loss in the first twelve months after laparoscopic Roux-en-Y gastric bypass (LRYGB).

Study design: Double-blind randomized placebo-controlled intervention study

Study population: Patients undergoing LRYGB at the bariatric expertise center for obesity of the Maasstad Hospital Rotterdam.

Intervention and procedure: Inclusion will take place at the outpatient clinic of the bariatric expertise center for obesity of the Maasstad Hospital. Patients will be randomly assigned to either the intervention or control group before surgery. The intervention group will receive a clear protein powder shake of 200 ml containing 20 grams of whey protein which should be taken daily during the first six months after LRYGB. The control group will receive an isocaloric, clear, placebo shake containing maltodextrine.

Main study parameters/endpoints: The main study parameter is the percentage fat free mass loss six months after surgery, calculated as fat free mass loss (kg) divided by total weight loss (kg) x 100%. Fat free mass will be assessed by multi-frequency bioelectrical impedance analysis (MF-BIA). Secondary parameters are percentage fat free mass loss, total weight loss, fat mass loss, BMI, hand grip strength, total protein intake and its progression over time, measured at baseline, 3, 6 and 12 months of follow-up.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: No additional outpatient visits will be required for study participants. A three day food diary and physical activity questionnaire must be filled out by all study participants at five regular follow-up moments. Body composition and handgrip strength will be assessed during these visits. All study participants will be asked to drink a daily shake, either protein or placebo, integrated in their postoperative diet. Study participants will receive information about the changes in body composition after surgery which is considered to be a significant benefit for patients participating in this study. The risk of participation is considered low. The risk consists of a possible allergic reaction to either the protein shake or the placebo.

ELIGIBILITY:
Inclusion Criteria:

* - Scheduled for a laparoscopic Roux-en-Y Gastric Bypass
* Age 18 - 65 years
* Body Mass Index ≥ 35 with the presence of severe comorbidity related to morbid obesity (diabetes mellitus type 2, obstructive sleep apnoea syndrome (OSAS), hypertension, etc.) or a BMI ≥ 40 with or without the presence of severe comorbidity related to morbid obesity
* Written informed consent

Exclusion Criteria:

* - Revisional bariatric surgery
* A protein-restricted diet for medical reasons
* Diagnosis of a (neuro-) muscular disease
* Inability to undergo MF-BIA (i.e. pregnancy, pacemaker)
* Allergy to any of the ingredients of either the protein or the placebo shake

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Fat Free mass loss | Change of fat free mass at 6 months post surgery compared to pre surgery
  Main study endpoint is percentage fat free mass loss at 6 months defined as fat free mass loss (kg) divided by total weight loss (kg) x 100%. Fat free mass will be assessed using the Seca® MBCA 515, which is a multi-frequency bio-electrical impedance analysis (MF-BIA). MF-BIA is an easy and non-invasive measurement tool and has been validated in morbid obese patients (13, 14). BIA measurements will be conducted under standardized circumstances. Patients can wear light clothes, have to empty their pockets and have to have an empty bladder. Patients will be asked to have no intensive physical activity and to have no food and fluid intake two hours prior to the measurements to minimalize bias.

SECONDARY OUTCOMES:
percentage of fat free mass loss, | Change of percentage fat free mass at 6 months post surgery compared to pre surgery
  measured by BIA
total weight loss, | pre surgery, 1 month after surgery, 3 months after surgery, 6 months after surgery, 12 months after surgery
  measured by BIA
fat mass loss, | Change of fat mass at 6 months post surgery compared to pre surgery
  measured by BIA
BMI | Change of BMI at 6 months post surgery compared to pre surgery
  measured by BIA
hand grip strength, | Change of hand grip strength at 6 months post surgery compared to pre surgery
  measured by hand grip strength device
total protein intake | Change of total protein intake at 6 months post surgery compared to pre surgery
  measured by 3 day food diary

CONTACTS AND LOCATIONS:
Overall Officials: Klaassen, MD, Principal Investigator — Maasstad Hospital
Locations (1):
- Maasstad Hospital, Rotterdam, South Holland, Netherlands

REFERENCES:
- [Derived] Taselaar AE, Boes AJ, de Bruin RWF, Kuijper TM, Van Lancker K, van der Harst E, Klaassen RA. PROMISE: effect of protein supplementation on fat-free mass preservation after bariatric surgery, a randomized double-blind placebo-controlled trial. Trials. 2023 Nov 9;24(1):717. doi: 10.1186/s13063-023-07654-w. PMID 37946272